CLINICAL TRIAL: NCT01618214
Title: A 20-week, Randomised, Open-label, 2-armed, Parallel Group Comparison of Subject-driven Titration of Biphasic Insulin Aspart (BIAsp) 30 Twice Daily Versus Investigator-driven Titration of BIAsp 30 Twice Daily Both in Combination With Oral Antidiabetic Drugs in Subjects With Type 2 Diabetes Inadequately Controlled With Premixed Human Insulin
Brief Title: Comparison of Subject-driven Titration of Biphasic Insulin Aspart (BIAsp) 30 Twice Daily Versus Investigator-driven Titration of BIAsp 30 Twice Daily Both in Combination With Oral Antidiabetic Drugs in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-3984; U1111-1126-7610 (Other: WHO)
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Results first posted 2014-05-08 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subject-driven titration (Experimental)
  Interventions: Drug: biphasic insulin aspart 30
- Investigator-driven titration (Active Comparator)
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Dose individually adjusted, administered subcutaneously (s.c., under the skin) twice daily.

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to compare BIAsp 30 twice daily individually adjusted by the subject versus BIAsp 30 twice daily individually adjusted by the investigator both combined with oral antidiabetic drugs (OADs) in subjects with type 2 diabetes inadequately controlled with premixed human insulin. Subjects to continue their OAD background treatment: Metformin plus/minus alpha-glucosidase inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Type 2 diabetes mellitus (diagnosed clinically) for at least 12 months
* Currently treated with premixed/self-mixed human insulin (proportion of short-acting insulin is equal to or lower than 30%) BID (twice daily) combined with metformin with or without alpha-glucosidase inhibitor for at least 3 months prior to screening visit (Visit 1) with the minimum dose stated: Metformin: at least 1500 mg/day or maximum tolerated dose at least 1000 mg/day (with unchanged dosing within 3 months prior to Visit 1) OR alpha-glucosidase inhibitors: acarbose or miglitol at least 150 mg/day, or voglibose at least 0.6 mg/day
* Total daily insulin dose below 1.4 IU/Kg
* HbA1c above or equal to 7.0% and below or equal to 9.5% (central laboratory)
* Body Mass Index (BMI) below or equal to 35.0 kg/m^2

Exclusion Criteria:

* Treatment with any insulin secretagogue, thiazolidinedione (TZD), dipeptidyl peptidase-4 (DPP-4) inhibitors and Glucagon-like peptide-1 (GLP-1) receptor agonists within the last 3 months prior to Visit 1
* Previous use of insulin intensification treatment (premixed insulin thrice daily, basal bolus regimen, and continuous subcutaneous insulin infusion (CSII)) for more than 14 days
* Previous use of any insulin other than premixed/self-mixed human insulin (proportion of short acting insulin equal to or lower than 30%) BID within 3 month prior to Visit 1
* Recurrent severe hypoglycaemia (more than 1 severe hypoglycaemic episode, during the last 12 months) or hypoglycaemic unawareness as judged by the investigator or hospitalisation for diabetic ketoacidosis during the previous 6 months
* Known proliferative retinopathy or maculopathy requiring treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2012-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (16):
- China (16):
  - Novo Nordisk Investigational Site, Hefei, Anhui
  - Novo Nordisk Investigational Site, Beijing, Beijing Municipality
  - Novo Nordisk Investigational Site, Chongqing, Chongqing Municipality
  - Novo Nordisk Investigational Site, Guangzhou, Guangdong
  - Novo Nordisk Investigational Site, Shijiazhuang, Hebei
  - Novo Nordisk Investigational Site, Wuhan, Hubei
  - Novo Nordisk Investigational Site, Tongliao, Inner Mongolia
  - Novo Nordisk Investigational Site, Nanjing, Jiangsu
  - Novo Nordisk Investigational Site, Yangzhou, Jiangsu
  - Novo Nordisk Investigational Site, Nanchang, Jiangxi
  - Novo Nordisk Investigational Site, Changchun, Jilin
  - Novo Nordisk Investigational Site, Siping, Jilin
  - Novo Nordisk Investigational Site, Xi'an, Shaanxi
  - Novo Nordisk Investigational Site, Jinan, Shandong
  - Novo Nordisk Investigational Site, Shanghai, Shanghai Municipality
  - Novo Nordisk Investigational Site, Hangzhou, Zhejiang

REFERENCES:
- [Result] Yang W, Zhu L, Meng B, Liu Y, Wang W, Ye S, Sun L, Miao H, Guo L, Wang Z, Lv X, Li Q, Ji Q, Zhao W, Yang G. Subject-driven titration of biphasic insulin aspart 30 twice daily is non-inferior to investigator-driven titration in Chinese patients with type 2 diabetes inadequately controlled with premixed human insulin: A randomized, open-label, parallel-group, multicenter trial. J Diabetes Investig. 2016 Jan;7(1):85-93. doi: 10.1111/jdi.12364. Epub 2015 May 25. PMID 26816605
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 23 sites in 1 country.
Pre-assignment Details: Eligible subjects were randomised in a 1:1 manner to one of the 2 treatment groups.
Groups:
- Subject-driven Titration: Subjects were transferred on a 1:1 basis from pre-trial premixed/self-mixed human insulin to biphasic insulin aspart 30 (BIAsp 30). Individually adjusted BIAsp 30 was given immediately before breakfast and dinner during 20 weeks. Subjects were trained on how to adjust BIAsp 30 doses during the training period [4 weeks] and then were asked to adjust their BIAsp 30 doses by themselves during the maintenance period [16 weeks]. Subjects continued their pre-trial oral anti-diabetic drugs (OADs) (metformin and/or alpha-glucosidase inhibitor). OADs were kept unchanged in regimen and daily dose during this trial, and were administered orally according to local labels.
- Investigator-driven Titration: Subjects were transferred on a 1:1 basis from pre-trial premixed/self-mixed human insulin to biphasic insulin aspart 30 (BIAsp 30). Individually adjusted BIAsp 30 was given immediately before breakfast and dinner during 20 weeks. Subjects were asked to adjust their BIAsp 30 doses according to the directions from investigators throughout the trial period [20 weeks]. Subjects continued their pre-trial oral anti-diabetic drugs (OADs) (metformin and/or alpha-glucosidase inhibitor). OADs were kept unchanged in regimen and daily dose during this trial, and were administered orally according to local labels.
Period: Overall Study
Arm/Group | Subject-driven Titration | Investigator-driven Titration
Started | 172 | 172
Exposed | 172 | 172
Completed | 162 | 159
Not Completed | 10 | 13
Not completed — Adverse Event | 3 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — Protocol Violation | 1 | 4
Not completed — Withdrawal Criteria | 1 | 2
Not completed — Unclassified | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subject-driven Titration | Investigator-driven Titration | Total
Number analyzed (Participants) | 172 | 172 | 344
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (7.3) | 53.4 (7.5) | 54.1 (7.4)
Gender [Count of Participants; unit: Participants]
  Female | 79 | 101 | 180
  Male | 93 | 71 | 164
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 172 | 172 | 344
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 70.3 (11.3) | 69.5 (11.6) | 69.9 (11.5)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.76 (3.26) | 25.47 (3.01) | 25.62 (3.14)
Glycosylated Haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.10 (0.64) | 8.14 (0.67) | 8.12 (0.65)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mmol/L] | 8.83 (2.36) | 9.07 (2.43) | 8.95 (2.40)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (Glycosylated Haemoglobin)
Description: Estimated mean change from baseline in HbA1c after 20 Weeks of treatment in full analysis set (FAS).
Time Frame: Week 0, week 20
Population: Full analysis set (FAS) - included all randomised subjects and missing data was imputed using last observation carried forward (LOCF) where any post-randomisation measurements were available. Six subjects did not contribute to FAS due to lack of post-randomisation measurements.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | Subject-driven Titration | Investigator-driven Titration
Number analyzed (Participants) | 168 | 170
percentage of glycosylated haemoglobin | -1.32 (0.86) | -1.31 (0.96)
Statistical Analysis 1: Comparison: Subject-driven Titration vs Investigator-driven Titration; FAS; Test type: Non-Inferiority or Equivalence — Non-inferiority was considered confirmed if the upper bound of the two-sided 95% confidence interval was below or equal to 0.4%; Regression, Linear; Mean Difference (Final Values) = -0.02, 95% CI [-0.19 to 0.14], Standard Deviation 0.08

2. Secondary Outcome: Percentage of Subjects Achieving HbA1c Below 7.0%
Time Frame: After 20 weeks of treatment
Population: Full analysis set (FAS) - included all randomized subjects and missing data was imputed using last observation carried forward (LOCF) where any post-randomization measurements were available.
Measure: Number; unit: percentage (%) of subjects
Arm/Group | Subject-driven Titration | Investigator-driven Titration
Number analyzed (Participants) | 172 | 172
percentage (%) of subjects | 64.5 | 58.1

3. Secondary Outcome: Percentage of Subjects Achieving HbA1c Below or Equal to 6.5%
Time Frame: After 20 weeks of treatment
Population: as for outcome 2
Measure: Number; unit: percentage (%) of subjects
Arm/Group | Subject-driven Titration | Investigator-driven Titration
Number analyzed (Participants) | 172 | 172
percentage (%) of subjects | 35.5 | 37.2

4. Secondary Outcome: Change From Baseline in FPG (Fasting Plasma Glucose)
Time Frame: Week 0, week 20
Population: Full analysis set (FAS) - included all randomized subjects and missing data was imputed using last observation carried forward (LOCF) where any post-randomization measurements were available. Seven subjects did not contribute to FAS due to lack of post-randomization measurements.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Subject-driven Titration | Investigator-driven Titration
Number analyzed (Participants) | 168 | 169
mmol/L | -1.26 (2.59) | -1.48 (3.01)

5. Secondary Outcome: Incidence of Hypoglycaemic Episodes (All, Major, Minor and Symptoms Only)
Description: Definition of a treatment emergent hypoglycemic episode: an episode occurred after the first administration of insulin or oral anti-diabetic drug, and no later than the last day on trial product. Severe hypoglycemic episode was that requiring assistance to administer carbohydrate, glucagon, or other resusciative actions. Minor hypoglycemic episode was the one with plasma glucose value < 3.1 mmol/L, either with symptoms that could be handled by subject, or without symptoms.
Time Frame: Week 0 to week 20 (inclusive).
Population: Safety Analysis Set (SAS) included all subjects receiving at least one dose of biphasic insulin aspart 30.
Measure: Number; unit: events per patient per year
Arm/Group | Subject-driven Titration | Investigator-driven Titration
Number analyzed (Participants) | 172 | 172
events per patient per year
  All hypoglycemic events | 10.04 | 10.90
  Severe hypoglycemic events | 0.02 | 0.02
  Minor hypoglycemic events | 1.70 | 1.66
  Probable symptomatic hypoglycemia | 0.45 | 0.56

ADVERSE EVENTS:
Time Frame: The reported treatment emergent adverse event was defined as an event that had onset date on or after the first day of exposure to randomised treatment and no later than the last day of randomised treatment, up to 20 weeks.
Description: Safety Analysis Set (SAS) included all subjects receiving at least one dose of biphasic insulin aspart 30.
Arm/Group | Subject-driven Titration | Investigator-driven Titration
Serious Adverse Events (participants affected / at risk) | 4/172 | 7/172
Other Adverse Events (participants affected / at risk) | 1/172 | 13/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subject-driven Titration (N=172) | Investigator-driven Titration (N=172)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Meniere (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) — All adverse events were coded using the Medical Dictionary for Regulatory Activities (MedDRA15.1).
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heat Stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenosquamous cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subject-driven Titration (N=172) | Investigator-driven Titration (N=172)
Influenza (Infections and infestations) | 1 (1) | 13 (15) — All adverse events were coded using the Medical Dictionary for Regulatory Activities (MedDRA15.1).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Novo Nordisk reserves the right to prior review of such publications and to ask for delay of publication of individual site results until after the primary manuscript is accepted for publication.